CLINICAL TRIAL: NCT06266585
Title: Risk Factor Analysis and Development of a Predictive Model for Clinical Deterioration During Hospitalization in Patients With Cerebral Venous Thrombosis
Brief Title: Clinical Deterioration in Cerebral Venous Thrombosis: A Predictive Study
Status: Completed | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Beijing Chao Yang Hospital (Other); Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Wang Shuo, Director of Department of cerebrovascular Neurosurgery, Beijing Tiantan Hospital
Other Study IDs: HX-B-2023090
Record Dates: First submitted 2024-01-05; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Cerebral Venous Thrombosis
MeSH Terms: conditions — Intracranial Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this retrospective, prospective, multicenter cohort study is to determine the risk factors for deterioration of CVT patients after admission and establish a scoring model for risk stratification of patients. This study included two stages, the first stage was to enroll CVT patients from a single center from 2017 to 2022 for modeling, and the second stage was to enroll CVT patients from three centers in 2023 for external validation

ELIGIBILITY:
Inclusion Criteria:

* Age≥ 18 years old
* Patients were diagnosed with cerebral venous thrombosis (CVT) through imaging techniques such as Computed Tomography Venography (CTV), Magnetic Resonance Venography (MRV), or Digital Subtraction Angiography (DSA)
* The diagnostic algorithm for CVT conformed to the current guideline criteria

Exclusion Criteria:

* Patients who had performed endovascular treatment (EVT) or decompressive craniectomy (DC) before admission and those whose primary treatment was EVT or DC rather than conservative treatment after admission
* Patients with severe hepatic or renal insufficiency
* Patients with intracranial tumors
* Patients with other cerebrovascular diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cerebral venous thrombosis (CVT)
Sampling Method: Non-Probability Sample
Enrollment: 273 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with CVT deteriorated on radiology | After admission until discharge, a maximum of 30 days
  One of the following situations occurs: new or progressive bleeding or infarction, midline displacement (>3mm), increased cerebral edema, and placeholder effect by comparing the CT before and after; mRS and/or GCS decreased due to decreased consciousness, increased focal neurological impairment, new focal neurological impairment or death.
Number of Participants with altered neurological function | After admission until discharge, a maximum of 30 days
  mRS Score decreased due to decreased consciousness, increased focal neurological impairment, new focal neurological impairment or death.
Number of Participants with altered consciousness | After admission until discharge, a maximum of 30 days
  GCS Score decreased

SECONDARY OUTCOMES:
Neurological function at 30th day after onset (mRS) | 30th day after onset
  MRS was used to evaluate the neurological function of patients at 30th day after onset.
Emergency surgery rates | After admission until discharge, a maximum of 30 days
  Rate of patients receiving emergency surgery for severe brain edema or hernia (including endovascular treatment and bone flap decompression).

CONTACTS AND LOCATIONS:
Locations (1):
- Capital Medical University Affiliated Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Feng Y, Mo S, Li X, Jiang P, Wu J, Li J, Liu P, Wang S, Liu Q, Tong X. Development and validation of a score for clinical deterioration in patients with cerebral venous thrombosis. Neurosurg Rev. 2025 Jan 16;48(1):56. doi: 10.1007/s10143-025-03224-7. PMID 39815140